CLINICAL TRIAL: NCT06876038
Title: A Comprehensive Platform for Low-cost Screening and Image-guided Photodynamic Therapy (PDT) Treatment of Pre-malignant and Malignant Oral Lesions in Low-resource Setting
Brief Title: Low-cost Screening and Image-guided Photodynamic Therapy (PDT) of Premalignant and Malignant Oral Lesions
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Massachusetts, Boston (Other)
Collaborators: Massachusetts General Hospital (Other); University of Arizona (Other); Aligarh Muslim University (Other); Karkinos Healthcare Hospitals Ernakulam, Kerala, India (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jonathan Celli, Professor, University of Massachusetts, Boston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA279862; U01CA279862 (NIH)
Record Dates: First submitted 2025-03-09; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-01

CONDITIONS: Oral Cancer; Oral Cavity Cancer; Oral Leukoplakia; Oral Lichen Planus; Oral Squamous Cell Carcinoma
Keywords: High grade dysplasia (HGD); Severe/Moderate dysplasia; Carcinoma-in-situ (CIS); Oral potentially malignant lesion (OPML)
MeSH Terms: conditions — Mouth Neoplasms; Leukoplakia, Oral; Lichen Planus, Oral; Squamous Cell Carcinoma of Head and Neck; Carcinoma in Situ | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- To evaluate the clinical efficacy of image guided photodynamic therapy to manage HGD-OPML (Experimental): The participants will take 5-ALA in oral solution (20 mg/kg BW 5-ALA HCl) 2 to 4 hours prior to undergoing image guided SITOS based PDT treatment. PDT treatment will use a total light dose of 100 J/cm^2 of 635 nm light (red light) delivered from a laser at an irradiance of approximately 50 mW/cm^2 at the tissue surface. Participants will be admitted for 48 hours to monitor toxicity profile evaluation. The lesion response will be evaluated and the PDT treatment will be repeated, if required, once in every 3 weeks with a maximum of up to three sessions. The clinical responses will be evaluated during the clinical visits. If the patient shows complete clinical response in less than three sessions of PDT, the PDT will be stopped and the patients will be followed up every 3 months, for one year. If there is lack of complete response or relapse of the lesions during the follow up, the patients will be advised to undergo surgical excision.
  Interventions: Drug: 5-Amino Levulinic Acid

INTERVENTIONS:
Drug: 5-Amino Levulinic Acid — 5-ALA (Gleolan) orally (20 mg/kg BW 5-ALA HCl) 2 to 4 hours prior to undergoing image-guided SITOS-based PDT treatment
  Other Names: Gleolan

SUMMARY:
The primary goal of this study is to see if photodynamic therapy (PDT) is effective for treatment of lesions in the oral cavity which have high risk of becoming oral cancer. PDT treatment uses a drug, called a photosensitizer, which makes the diseased cells become light-sensitive such that they are destroyed when laser light is delivered to the target lesion. In this study a new handheld device, called SITOS (a "Screen, Image and Treat Optical System), is used. The ability of this device to simultaneously visualize the inside of the mouth and deliver laser light to the target site will be evaluated. The main questions this study seeks to answer are:

* Can this treatment completely cure oral potentially malignant lesions (OPML) without need for surgery?
* Do lesions recur after PDT treatment?
* Is the SITOS device easy to use for the doctor and comfortable for the patient, both as an oral imaging device and as a treatment device?

DETAILED DESCRIPTION:
This study seeks to evaluate the efficacy of photodynamic therapy (PDT) using aminolevulinic acid (ALA) photosensitization for treatment of oral potentially malignant lesions (OPML) or early stage oral cancer. Eligible participants will have histopathologically confirmed high-grade dysplasia/HGD (severe/moderate dysplasia) or early stage cancer (carcinoma-in-situ, CIS) in the oral cavity. While PDT using ALA photosensitization has already been shown to be safe and effective for other indications it is not yet approved for use in treatment of oral lesions. Preliminary clinical studies have indicated that PDT is well tolerated and can achieve complete clearance of lesions with excellent healing of the oral mucosa. This study specifically seeks to evaluate the use of a new handheld optical device called the Screen, Image, and Treat Optical System (SITOS) which combines imaging and PDT light delivery. This device, which is similar in size and shape to a standard dental camera, contains integrated optics for imaging the characteristic fluorescence signal which results from ALA-induced protoporpohpryin IX photosensitization. This will be used for imaging-based guidance of light delivery for PDT, which uses a red diode laser that is also integrated into the device.

Potential study participants will be identified in screening sessions at the participating clinical sites or through referral. Those with potentially qualifying lesions and who consent to participate undergo will undergo pre-treatment investigation, including clinical information on the oral lesion, risk profile and baseline toxicity profile, and preliminary imaging.

For those who qualify for PDT treatment, photosensitization will use 5-ALA (20 mg/kg body weight 5-ALA-HCl, Gleolan) administered orally 2 to 4 hours before treatment. After administration of 5-ALA, exposure of eyes and skin to strong light sources (e.g., operating illumination, direct sunlight, or brightly focused indoor light) must be avoided for 24 hours. The lesion area to be treated will be anesthetized locally with 2% xylocaine with 1:100,000 adrenalin. If the patient or the investigator desires, he/she may undergo the procedure under general anesthesia or IV sedation. Following administration of 5-ALA, the participant will undergo image-guided SITOS-based PDT treatment. SITOS will be used in the imaging mode to establish background fluorescence before 5-ALA administration, and again after ALA photosensitization to provide visualization of the photosensitized lesion. For photoactivation, a total light dose of 100 J/cm^2 will require ~30 minutes, depending on the final irradiance generated by SITOS. This may be given in 10-minute fractions with brief breaks for comfort. At light delivery time, SITOS will be used for real-time visualization of light applicator positioning to ensure centering of the beam spot and margins around the lesion. The SITOS probe also has a snap-on collar to control spacing and beam spot size which is fixed in place. A bitewing is clipped on for stable positioning with a hygienic sleeve over the whole probe. SITOS will monitor photobleaching (the decrease in fluorescence due to photosensitizer degradation during PDT) in real time, switching to image mode with brief interruptions in light delivery (approximately ~ 1 sec). Once per minute, measurement of bleaching relative to pre-irradiation will be performed. Participants will be kept in a room without direct sunlight exposure. The patients will be discharged after 48 hours of monitoring and toxicity profile evaluation.

The lesion response will be evaluated three weeks after PDT treatment. If complete response is not observed PDT may be repeated for a maximum of three sessions total. The clinical responses will be defined as complete, partial, and not responding as per the modified RECIST criteria. The final response will be determined in three weeks after the last PDT treatment (maximum of three sessions). If the patients show complete clinical response in less than three sessions of PDT, the PDT will be stopped, and the patients will be followed up every 3 months for one year. Punch biopsy will be performed to confirm histologic response a minimum of three months after the last PDT administration. Any lesions showing histologic evidence of dysplasia are considered a persistent disease and recommended to undergo surgical excision.

ELIGIBILITY:
Subject Inclusion Criteria

1. One grossly visible OPML, with histopathologically confirmed diagnosis of moderate, severe, and carcinoma in situ measuring ≥ 10 mm in diameter.
2. Willing and available for follow-up for at least one year and at prerequisite time intervals.
3. All patients above the age of 18 years and willing to voluntarily give a signed informed consent.
4. Karnofsky Performance Score above 80 or ECOG 0 or 1.
5. The subjects meeting the following laboratory eligibility criteria during a time not older than 2 months before accrual

   * Hemoglobin level above or equal to 10%
   * WBC >3000/mm3
   * Platelets count >100000/mm3
   * Total bilirubin, AST (SGOT), ALT (SGPT) < 1.5 times the Upper Limit Normal
   * eGFR > 60 ml/min
   * Serum Creatine less than 2 times the Upper Limit of laboratory normal
   * INR/ PT and PTT within laboratory normal limits

Exclusion criteria:

1. Hypersensitivity against active substances and porphyrins.
2. Known diagnosis of porphyria.
3. Simultaneous use of other potentially phototoxic substances (eg; tetracyclines, sulphonamides, fluoroquinolones, hypericin extracts).
4. Uncontrolled concurrent illness, including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled cardiac and renal diseases or psychiatric illness.
5. Subjects with inherited or acquired bleeding and clotting disorders
6. Women who are breastfeeding/ have a positive urine pregnancy test or are planning their family.
7. Patients who have taken supplements of retinol, beta carotene, vitamin E, Selenium, or other chemo-preventive therapy at least one month prior to the baseline visit.
8. Patients with histological evidence of no dysplasia, mild dysplasia, invasive carcinoma, and any active malignant disease.
9. Patients with behavioral and cognitive impairment.
10. Patients who are concurrently diagnosed and undergoing treatment for other head and neck cancers.
11. Patients with large lesions, which, in the investigator's opinion, may require reconstructive surgery after excision.
12. The subjects, in the opinion of the Institutional Principal Investigator, are not an appropriate candidate for study participation due to alcoholism and abstinence.
13. Patient who was in a clinical trial for 4 weeks before participation in the present trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy of 5-ALA based PDT to treat HGD-OPML | 3 weeks after PDT treatment
  The response will be clinically evaluated three weeks after PDT treatment. It will be defined as complete, partial, stable or progressive disease by modified RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Tayyaba Hasan, PhD, Principal Investigator — Massachusetts General Hospital, Boston, MA, United States; Jonathan Celli, PhD, Principal Investigator — University of Massachusetts Boston, Boston, MA, United States; Moni A Kuriakose, MD, Principal Investigator — Karkinos Healthcare Hospitals Ernakulam, Kerala, India; Mohammad Akram, MD, Principal Investigator — Aligarh Muslim University, Aligarh, Uttar Pradesh, India
Locations (2):
- India (2):
  - Karkinos Healthcare Hospitals, Ernākulam, Kerala
  - Jawaharlal Nehru Medical College, AMU, Aligarh, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified clinical data which underlie published results will be available for sharing as per requirements of the journal in which study results are reported.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available in compliance with publishers data availability policy, starting from the date of publication.
Access Criteria: A data sharing agreement must first be established between the requester and the study team and their respective institutional officials. Data eligible for sharing will include any raw data that directly underlies published results (clinical reports, raw images and statistical analyses). Once a data sharing agreement is established the data can be shared using a secure link to a shared OneDrive folder or other appropriate and secure file sharing platform.

REFERENCES:
- [Background] Siddiqui SA, Siddiqui S, Hussain MAB, Khan S, Liu H, Akhtar K, Hasan SA, Ahmed I, Mallidi S, Khan AP, Cuckov F, Hopper C, Bown S, Celli JP, Hasan T. Clinical evaluation of a mobile, low-cost system for fluorescence guided photodynamic therapy of early oral cancer in India. Photodiagnosis Photodyn Ther. 2022 Jun;38:102843. doi: 10.1016/j.pdpdt.2022.102843. Epub 2022 Mar 31. PMID 35367616